CLINICAL TRIAL: NCT05745207
Title: A First-In-Human, Two-Part Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2086 in Healthy Adult and Elderly Subjects
Brief Title: A Study To Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2086 in Healthy Adult and Elderly Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: E2086-A001-001
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A, Cohort 1: E2086 1 mg or Placebo (Experimental): Participants will receive 1 milligram (mg) (2*0.5 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo
- Part A, Cohort 2: E2086 2.5 mg or Placebo (Experimental): Participants will receive 2.5 mg (5*0.5 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo
- Part A, Cohort 3: E2086 5 mg or Placebo (Experimental): Participants will receive 5 mg (1*5 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo
- Part A, Cohort 4: E2086 10 mg or Placebo (Experimental): Participants will receive 10 mg (2*5 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo
- Part A, Cohort 5: E2086 25 mg or Placebo (Experimental): Participants will receive 25 mg (1*25 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo
- Part A, Cohort 6: E2086 50 mg or Placebo (Experimental): Participants will receive 50 mg (2*25 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo
- Part A, Cohort 7: E2086 100 mg or Placebo (Experimental): Participants will receive 100 mg (4*25 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo
- Part B, Cohort 8: E2086 25 mg or Placebo (Experimental): Participants will receive 25 mg (1*25 mg) E2086 or E2086 matched placebo, tablets, orally, once on Day 1.
  Interventions: Drug: E2086; Drug: Placebo

INTERVENTIONS:
Drug: E2086 — E2086 tablets.
Drug: Placebo — E2086 matched placebo tablets.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of E2086 following administration of a single oral doses in healthy adult and elderly participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, male or female, age greater than or equal to (>=) 18 years to less than or equal to (<=) 55 years old (greater than [>] 65 years old for Part B) at the time of informed consent. To be considered non-smokers, participants must have discontinued smoking for at least 4 weeks before dosing.
2. Reports regular bedtime, defined as the time the participant attempts to sleep, between 21:00 and midnight, based on sleep diary data from the Screening Period.
3. Reports regular waketime, defined as the time the participant gets out of bed for the day, between 05:00 and 10:00, based on sleep diary data from the Screening Period.
4. Body mass index (BMI) >=18 to less than (<) 30 kilogram per square meter (kg/m^2) at Screening.

Exclusion Criteria:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 international units per liter (IU/L) or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the dose of study drug.
3. All females who are of childbearing potential:

   • All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
4. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period or for 90 days after study drug discontinuation
5. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing (example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system)
6. Any history of a congenital abnormality in metabolism at Screening
7. Any history of seizure, epilepsy, or non-epileptic seizures
8. Any history of surgery that may affect PK profiles of E2086 (example, hepatectomy, nephrotomy, digestive organ resection) at Screening
9. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening or Baseline
10. Liver function test values outside of the normal laboratory defined range at Screening or Baseline.
11. Any history of liver disease.
12. Known history of liver function test values outside of the normal laboratory defined range within the last 6 months.
13. Evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease, sleep disorders) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
14. A prolonged QT/QTc interval (QTc >450 milliseconds [ms]) demonstrated on ECG at Screening or Baseline (based on average of triplicate ECGs). A history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
15. Left bundle branch block at Screening or Baseline
16. Persistent systolic BP >130 or <100 millimeters of mercury (mmHg) or diastolic BP >85 or <50 mmHg at Screening or Baseline (based on BP measured on at least 3 occasions over 2 weeks)
17. Persistent heart rate (HR) less than 50 beats/min or more than 100 beats/min at Screening or Baseline (based on HR measured on at least 3 occasions over 2 weeks)
18. History of myocardial infarction, ischemic heart disease, or cardiac failure at Screening
19. History of clinically significant arrhythmia or uncontrolled arrhythmia
20. Known history of clinically significant drug allergy at Screening or Baseline
21. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
22. Known to be human immunodeficiency virus (HIV) positive at Screening
23. Active or chronic viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
24. Active Epstein Barr virus (EBV) as demonstrated by positive serology at Screening
25. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive drug test or alcohol test at Screening or Baseline
26. Intake of caffeinated beverages or food within 72 hours before dosing
27. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing
28. Any lifetime history of suicidal ideation or any lifetime history of suicidal behaviour as indicated by the Columbia-Suicide Severity Rating Scale (C-SSRS).
29. Any lifetime history of psychiatric disease (including but not limited to depression or other mood disorders, bipolar disorder, psychotic disorders, including schizophrenia, panic attacks, anxiety disorders). The absence of a history of psychiatric disease should be documented by a checklist in the eCRF.
30. Any current psychiatric symptoms as indicated by a standard screening tool (Diagnostic and Statistical Manual of Mental Disorders [DSM-5] Self-Rated Level 1 Cross-Cutting Symptom Measure - Adult)
31. Participants who's 1st degree (blood) relatives have lifetime diagnosis of bipolar type I disorder or a psychotic disorder.
32. Use of prescription drugs within 4 weeks before dosing
33. Intake of over the counter (OTC) medications within 2 weeks before dosing
34. Currently enrolled in another clinical study or used any investigational drug or device within 30 days or 5 half-lives, whichever is longer, preceding informed consent
35. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing
36. Epileptiform discharges on screening EEG
37. History of formally diagnosed moderate to severe obstructive sleep apnea, current use of continuous positive airway pressure, or symptomatic restless legs syndrome.
38. Exposure within the last 14 days to an individual with confirmed or probable COVID-19 or symptoms within the last 14 days that are on the most recent Centers for Disease Control and Prevention (CDC) list of COVID symptoms or any other reason to consider the participant at potential risk for COVID-19 infection.
39. Exposure to any biologic drug within 90 days or at least 5 half-lives (whichever is longer), or within 4 weeks for vaccines, before Screening, with the exception of flu (7 days before dosing) and COVID-19 vaccination (14 days before dosing until after the Follow-up visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From Screening up to 10 days
Number of Participants With Serious Adverse Events (SAEs) | From Screening up to 10 days
Number of Participants With Clinically Significant Abnormal Laboratory Values | From Screening up to 10 days
Number of Participants With Clinically Significant Abnormal Vital Signs Values | From Screening up to 10 days
Number of Participants With Clinically Significant Abnormal Electrocardiograms (ECGs) Findings | From Screening up to 10 days
Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-suicide Severity Rating Scale (C-SSRS) | From Screening up to 10 days
  The C-SSRS is an interview-based rating scale to systematically assess any suicidality, suicidal behavior, or suicidal ideation. Any suicidality is emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior is indicated when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation is indicated when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.
Number of Participants With Clinically Significant Abnormal Physical Examination Findings | From Screening up to 10 days
Number of Participants With Clinically Significant Abnormal Neurological Examination Findings | From Screening up to 10 days
Number of Participants With Clinically Significant Abnormal Electroencephalogram (EEG) Findings | Baseline, Days 1 and 2

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
Tmax: Time to Reach Maximum Observed Plasma Concentration (Cmax) for E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
AUC(0-24h): Area Under the Plasma Concentration-time Curve From Time Zero to 24 hours Post-dose for E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 24 hours post-dose
AUC(0-t): Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration for E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
AUC(0-72h): Area Under the Plasma Concentration-time Curve From Time Zero to 72 hours Post-dose for E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 72 hours post-dose
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time Zero to Infinite for E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
t1/2: Terminal Elimination Phase Half-life for E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
CL/F: Apparent Total Clearance for E2086 | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
Vz/F: Apparent Volume of Distribution at Terminal Phase for E2086 | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
MRp: Ratio of Plasma AUC(0-inf) of Metabolite to E2082, Corrected for Molecular Weights | Day 1: Pre-dose (0 hour) up to 216 hours post-dose
Mean Change in Subjective Sleep Onset Latency (sSOL) | Screening up to Study Day 7
  sSOL is a participant-reported estimate of the amount of time (in minutes) it took the participant to fall asleep the prior evening.
Ae: Cumulative Amount of E2086 and its Metabolites Excreted in Urine | Day 1: Pre-dose (0 hour) up to 120 hours post-dose
CLR: Renal Clearance of E2086 and its Metabolites | Day 1: Pre-dose (0 hour) up to 120 hours post-dose
Fe: Percent (%) of E2086 and its Metabolites Excreted in Urine | Day 1: Pre-dose (0 hour) up to 120 hours post-dose
MRU: Ratio of Ae Urine Concentration of Metabolite to E2082, Corrected for Molecular Weights | Day 1: Pre-dose (0 hour) up to 120 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.